CLINICAL TRIAL: NCT00478452
Title: Randomized Phase I/II Pilot Study of the Immunogenicity of Cyclophosphamide With Peptide Pulsed Mature Dendritic Cells for Patients With Previously Treated Ovarian Epithelial or Primary Peritoneal Carcinoma
Brief Title: Dendritic Cell Vaccine for High Risk Ovarian Cancer Patients
Acronym: DC-Ova
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 707800; UPCC 01803 (Other: CTSRMC)
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to cyclophosphamide 300 mg/m2 (arm 2) or no cyclophosphamide (arm 1). All subjects will receive intradermal injections of DC on day 2 and on week 3, 6, and 9 (+ 3 days). All subjects will undergo leukocyte apheresis at study enrollment and at week 10, which is the end of active study intervention. All study arm patients (1 and 2) will receive a single dose of trivalent killed influenza vaccine, and a single dose of Prevnar pneumococcal vaccine on the day they receive their first intradermal injections of DC on day 2.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DC Ova (Experimental): DC Ova vaccine administered day 2 and week 3,6,9
  Interventions: Biological: DC-Ova
- DC Ova with Cyclophosphamide (Active Comparator): Cyclophosphomide administered at day 0 prior to administration of DC Ova vaccine administered day 2 and week 3,6,9
  Interventions: Biological: DC Ova with Cyclophosphamide

INTERVENTIONS:
Biological: DC-Ova
  Arms: DC Ova
Biological: DC Ova with Cyclophosphamide
  Arms: DC Ova with Cyclophosphamide

SUMMARY:
This is a randomized Phase I/II study designed to assess the induction of an anti-tumor immune response; the effect of cyclophosphamide on the vaccine; and to assess safety in subjects with advanced ovarian cancer or primary serous peritoneal cancer given a multivalent DC vaccine, with or without a single dose of cyclophosphamide.

Potential benefit may range from no direct benefit to the study participants to stimulation of the subject's own immune system to attack ovarian cancer to prevent relapse.

DETAILED DESCRIPTION:
HLA-A2+ subjects with stage II-IV who have completed chemotherapy and are in clinical remission or patients with stage I-IV advanced ovarian cancer or primary serous peritoneal cancer in clinical remission post treatment for disease recurrence occurring after a progression-free interval of at least two years will be eligible. Patients will be evaluated by standard imaging techniques. Patients will be randomized to cyclophosphamide 300 mg/m2 (arm 2) or no cyclophosphamide (arm 1). All subjects will receive intradermal injections of DC on day 2 and on week 3, 6, and 9 (+ 3 days). All subjects will undergo leukocyte apheresis at study enrollment and at week 10, which is the end of active study intervention. All study arm 1 and 2 patients (without prior vaccination with the current season's vaccine) will receive a single dose of trivalent killed influenza vaccine, and a single dose of Prevnar pneumococcal vaccine on the day they receive their first intradermal injections of DC on day 2.

ELIGIBILITY:
Inclusion Criteria:

* The following conditions must be met before a patient may be enrolled in the study.
* Patients age 18 years of age and older.

Disease Criteria. Patients will be eligible:

* If no clinical evidence of disease is present after diagnosis with stage III or
* IV disease and completion of primary surgery and chemotherapy, or, if no clinical evidence of disease is present after completion of chemotherapy for a disease recurrence diagnosed after a progression-free interval of at least 2 years, for patients of any initial stage.or primary peritoneal carcinoma.
* Complete clinical response = no evidence of tumor lesions shown by abdominal CT scan or MRI, chest Xray,and CA 125 level ≤ 35 UI/mL.
* Time from completion of Chemotherapy will be no more than 6 months from last dose from initial diagnoses.
* HLA-A2 positive (must be typed by molecular methods; all A2 alleles eligible).

Patients with adequate organ function as measured by:

* Hematopoietic: WBC at least 3000/mm3; platelets at least 100,000/mm3, hemoglobin at least 10.0 g/dL (may be transfused).
* Cardiac: Asymptomatic or, if symptomatic, then left ventricular ejection fraction at rest must be ≥50% or within the normal range of the institution. A cardiology clearance will be required for LV ejection fraction <50%.
* Hepatic: SGOT within 2x normal range and total bilirubin ≤ 2.0 mg/dL.
* Renal: Serum creatinine ≤2.0 mg/dL
* Adequate performance status > 80% (Karnofsky) or ECOG 0-2
* Written informed consent conforming to institutional guidelines.
* Life expectancy > 6 months and absence of co-existing medical problems which would preclude participation in the judgment of the principal investigator.

Exclusion Criteria:

* Any one of the following conditions eliminates a patient from participating in this protocol.
* Prior malignancy (except basal cell or squamous cell skin cancer) within the past five years.
* Presence of active Central Nervous System disease.
* Serious systemic disease.
* Active bacterial, viral or fungal infections.
* Chemotherapy, biologic therapy or radiation therapy less than 4 weeks prior to study entry.
* History of active autoimmunity or immunosuppression.
* Use of immunosuppressive drugs within 4 weeks prior to study entry or anticipated use of immunosuppressive agents.
* Patients with tumors of low malignant potential (borderline tumors) will not be eligible.
* Seropositivity for HIV, HTLV-1, or HTLV-2.
* Prior Influenza vaccination with the current vaccine will exclude patient from receiving protocol-specified influenza vaccine but will not exclude participation with the other aspects of the protocol. Each year's vaccine supply generally becomes available in October. Patients with a history of serious hypersensitivity to eggs, previous influenza vaccine or its components, will not receive influenza vaccine, but may continue to participate in other aspects of the protocol. Patients with a history of serious hypersensitivity to the Prevnar vaccine, its components, or diptheria toxoid will not receive the Prevnar vaccine, but may continue to participate in other aspects of the protocol.
* Pregnant or breast feeding subjects.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To assess the immunogenicity (with or without prior cyclophosphamide administration) of IDD-6, a peptide-loaded matured DC vaccine. | 24 months
  Immunogenicity will be assessed by determining the frequency of specific HLA A -restricted T cells following vaccination with her2/neu, hTERT and PADRE -loaded DC

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chu, MD, Principal Investigator — University of Pennsylvania Hospital
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: University of Pennsylvania Abramson Cancer Center Web Line — http://oncolink.com